CLINICAL TRIAL: NCT01354379
Title: A Phase 1 Randomized, Observer-Blind, Controlled, Safety, Tolerability and Immunogenicity Study of Intranasal NB-1008 in Healthy Adult Volunteers Administered by Nasal Sprayer and Pipette
Brief Title: Safety and Immunogenicity Study of Inactivated Nasal Influenza Vaccine NB-1008 Administered by Sprayer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NanoBio Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NB-1008-002
Record Dates: First submitted 2011-05-13; First posted 2011-05-16 (Estimated); Last update posted 2013-03-28 (Estimated); Status verified 2013-03

CONDITIONS: Healthy Adult Volunteers
MeSH Terms: interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Fluzone 15 mcg HA 200 mcl IN by Pipette (Active Comparator)
  Interventions: Biological: Fluzone IN
- NB-1008 15 mcg HA 20% W805EC 200 mcl IN by Pipette (Experimental)
  Interventions: Biological: NB-1008
- Fluzone 15 mcg HA 200 mcl IN by Nasal Spray (Active Comparator)
  Interventions: Biological: Fluzone IN
- NB-1008 15 mcg HA 20% W805EC 200 mcl IN by Nasal Spray (Experimental)
  Interventions: Biological: NB-1008
- NB-1008 15 mcg HA 20% W805EC 400 mcl IN by Nasal Spray (Experimental)
  Interventions: Biological: NB-1008

INTERVENTIONS:
Biological: NB-1008 — NB-1008 is composed of Fluzone containing 15 micrograms (mcg) of strain-specific hemagglutinin (HA) and 20% W805EC adjuvant.
  Arms: NB-1008 15 mcg HA 20% W805EC 200 mcl IN by Nasal Spray; NB-1008 15 mcg HA 20% W805EC 200 mcl IN by Pipette; NB-1008 15 mcg HA 20% W805EC 400 mcl IN by Nasal Spray
Biological: Fluzone IN — The active control is Fluzone containing 15 micrograms (mcg) of strain-specific hemagglutinin (HA).
  Arms: Fluzone 15 mcg HA 200 mcl IN by Nasal Spray; Fluzone 15 mcg HA 200 mcl IN by Pipette

SUMMARY:
The purpose of this study is to test the safety and immune response of a new intranasal vaccine against influenza, called NB-1008. The vaccine is composed of a licensed vaccine that is normally given as an injection, called Fluzone, and an adjuvant (additive that helps a vaccine work better), called W805EC. In a prior clinical study this vaccine showed promising results in terms of being well tolerated and eliciting mucosal and systemic immune responses after administration by a dropper. In this study NB-1008 is being administered by dropper as well as a nasal sprayer to determine if the sprayer further enhances the immune response.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female.
2. Are 18-49 years of age, inclusive.
3. If female, must be non-pregnant as confirmed by a negative serum pregnancy test conducted at screening and a negative urine pregnancy test conducted at the site within 24 hours preceding receipt of vaccine.
4. Females who are not surgically sterile or at least one year post-menopausal agree to use oral, implantable, transdermal or injectable contraceptive or another reliable form of contraception approved by the Investigator for a minimum of 30 days prior to vaccination and for 3 months following vaccination.
5. Healthy, as determined by medical history, physical examination, vital signs, and clinical laboratory examinations.
6. Comprehension of the study requirements, expressed availability for the required study period, and ability to attend scheduled visits.
7. Has given written informed consent to participate in the study.

Exclusion Criteria:

1. Presence of significant acute or chronic, uncontrolled medical or psychiatric illness (institution of new medical or surgical treatment, or a significant dose alteration for uncontrolled symptoms or drug toxicity within 3 months). Subjects with a history of chronic cough, frequent sinus infections, sinusitis, allergic rhinitis, nasal polyps or obstruction, including deviated septum significant enough to obstruct the nasal openings are to be excluded. Subjects with seasonal rhinitis may be included if their 'season' does not occur within 3 months of the vaccination date and they are not currently receiving intranasal steroids.
2. Receipt of the 22010-2011 influenza vaccine or the 2009 pandemic H1N1 influenza vaccine.
3. Positive serology for HIV-1 or HIV-2, or HCV antibodies.
4. Platelet count <150,000/mm3.
5. Positive urine drug screen.
6. History of aspiration, dysphagia, swallowing disorders, stroke or other neurologic conditions that may predispose the subject to aspiration of test articles into the respiratory tract.
7. History of Bell's palsy.
8. Cancer or treatment for cancer, within 3 years. Subjects with a history of cancer who are disease-free without treatment for 3 years or more are eligible. Basal cell carcinoma (BCC) or (SCC) are allowed, unless present on or near the nose.
9. Impaired immune responsiveness, regardless of cause, including diabetes mellitus.
10. Presently receiving or history of receiving any medications or treatments that affects the immune system such as immune globulin, interferon, immunomodulators, cytotoxic drugs or drugs known to be frequently associated with significant major organ toxicity, or systemic corticosteroids (oral or injectable) in the past 6 months.
11. Chronic use of inhaled or intranasal sprays including decongestants and corticosteroids.
12. Presently a smoker or tobacco user or have a history of smoking or tobacco use within the past year prior to screening.
13. Receipt or planned administration of a nonstudy vaccine within 30 days before the study, including licensed influenza vaccines and prior to the Day 60 telephone contact. Immunization on an emergency basis with Tetanus Toxoids Adsorbed for adult use (Td or Tdap) up to 8 days before or at least 8 days after a dose of study vaccine will be allowed. Administration of study vaccine can be delayed if a nonstudy vaccine has been administered and will be given as soon as acceptable, as described above.
14. Known allergy to any vaccine component, including eggs, egg products, or thimerosal.
15. History of allergic and/or anaphylactic type reaction to injected vaccines or to any of the components of NB-1008 [soybean oil, dehydrated alcohol (anhydrous ethanol), polysorbate (Tween 80) and cetylpyridinium chloride (CPC)].
16. History of drug or chemical abuse in the year before the study.
17. Receipt of any investigational product or nonregistered drug within the 30 days before study entry or currently enrolled in any investigational drug study or intends to enroll in such a study within the ensuing 6 month period.
18. Use of nasally administered prescription or over-the-counter (OTC) medications within 7 days before vaccination
19. Receipt of blood or blood products 8 weeks before study entry or planned administration prior to the Day 60 telephone contact.
20. Donation of blood or blood products within 8 weeks before study entry or at any time up to the Day 28 clinic visit.
21. Acute disease within a week prior to vaccination, defined as the presence of a moderate or severe illness (as determined by the investigator through medical history and physical examination) with or without fever. For subjects with a minor illness, such as diarrhea, or mild upper respiratory tract infection with or without low-grade febrile illness, the subject can be re-screened once they have complexly recovered.
22. Any condition that, in the opinion of the investigator, might interfere with study objectives.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2011-05; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | 365 Days
  Number of Participants with Adverse Events (AE) collected through Day 28 and Serious Adverse Events (SAE) collected through Day 365.

SECONDARY OUTCOMES:
Systemic Humoral Immune Response | Day 28 and Day 60
  Serum hemagglutination-inhibition (HAI) Geometric Mean Titer (GMT) and proportion of Volunteers with >=4 fold increase in titer as well as proportion of volunteers with titer >= protective level of 40
Systemic Cell Mediated Immune Response | Day 28
  Stimulation Index (SI) of antigen-specific proliferation and cytokine secretion of peripheral mononuclear cells (PBMC)
Mucosal Immune Response | Day 14 and Day 28
  Nasal wash anti-Fluzone IgA Geometric Mean Titer (GMT) and proportion of volunteers with >=4 fold increase in GMT anti-Fluuzone IgA titer

CONTACTS AND LOCATIONS:
Overall Officials: Casey T Johnson, DO, Principal Investigator — Johnson County Clin-Trials
Locations (1):
- Johnson County Clin-Trials, Lenexa, Kansas, United States